CLINICAL TRIAL: NCT06015503
Title: A Phase Ⅱ,Open-label, Single-line, Multiple Cohorts, Multicenter Study Assessing the Safety and Efficacy of PLB1004 in EGFR ex20ins Mutation Patients With Advanced and Metastatic Non-small Cell Lung Cancer(NSCLC)
Brief Title: A Phase Ⅱ Study Assessing the Safety and Efficacy of PLB1004 in EGFR ex20ins Mutation Patients With Advanced and Metastatic Non-small Cell Lung Cancer(NSCLC)
Acronym: KANNON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004-II-01
Record Dates: First submitted 2023-08-18; First posted 2023-08-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; EGFR; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PLB1004 (Experimental): PLB1004 given alone as monotherapy
  Interventions: Drug: PLB1004

INTERVENTIONS:
Drug: PLB1004 — PLB1004 is a capsule in the form of 80mg and 40mg.

SUMMARY:
It is a phase Ⅱ,open-label, single-line, Multiple cohorts, Multicenter study assessing the Safety and Efficacy of PLB1004 in EGFR ex20ins mutation patients with Advanced and Metastatic Non-small Cell Lung Cancer(NSCLC).

DETAILED DESCRIPTION:
This a three-stage study consist a Screening Phase (Day -28 to -1), a Treatment Phase (until treatment discontinuation), and a Follow-up Phase (including end of treatment visit (EOT),end of study visit(EOS), safety follow-up and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged at least 18 years old.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (stage IIIB~IV).
4. According to the prior treatments having received for advanced disease (platinum containing or/and immunotherapy containing systemic therapy, not more than three lines), participants were divided into two cohorts。
5. Participants with EGFR ex20ins mutation.
6. ECOG performance status 0 to 1.
7. Life expectancy is not less than 12 weeks.
8. At least one measurable lesion as defined by RECISTV1.1.
9. Participants must have specific organ and bone marrow function.

Exclusion Criteria:

* Exclusion

  1. Having the anticancer therapy prior to the first dose of PLB1004 as follows:

     1. Any monoclonal antibodies targeting EGFR/HER2/VEGFR within 4 weeks.
     2. Any cytotoxic drugs or other anticancer drugs from a previous treatment regimen within 14 days.
     3. Any anticancer herbal medicine within 7 days
     4. Major surgery within 4 weeks prior to starting PLB1004 or who have not recovered from side effects of such procedure except for the biopsy of Thoracoscopy and the clinical test of Mediastinoscopy could ≤ 7 days prior to starting PLB1004..
     5. Radiotherapy to lung fields and whole-brain fields ≤4 weeks prior to starting PLB1004. For all other anatomic sites, radiotherapy ≤2 weeks prior to starting PLB1004 or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions is not included.
     6. Any anti-EGFR TKI for the EGFR ex20ins mutation.
     7. Any third-generation anti-EGFR TKI during the treatment having achieved a best overall response of the partial response or complete response.
  2. Had not recovered from the adverse events and comorbidities caused by prior Systemic chemotherapy ,surgery ,radiotherapy to ≤ Grade 1（except for hair loss and permanent radiotherapy damage ）,the neurological toxicity caused by platinum could ≤ Grade 2.
  3. Patients receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with PLB1004 and for the duration of the study:

     * Strong inhibitors of CYP3A4
     * Strong inducers of CYP3A4
     * metformin a MATE transporter substrate
  4. Patients with spinal cord compression ,brain membrane metastasis and symptomatic central nervous system (CNS), who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study manage CNS symptoms.
  5. Patients with uncontrolled and symptomatic pleural effusions, peritoneal effusions and pericardial effusions within 4 weeks prior to the start of treatment with PLB1004.
  6. Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, indolent malignancies that currently do not require treatment, and completely resected carcinoma in situ of any type.
  7. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
  8. Konwn positive hepatitis B (hepatitis B virus , HBV) surface antigen(HBsAg) and HBV-DNA test value≥ULN.
  9. known positive hepatitis C antibody(anti-HCV) and Anti-HIV(+).Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
  10. Having significant or uncontrolled systemic disease, including but not limited to:

      1. Poorly controlled hypertension (referring to systolic blood pressure>100 mmHg after treatment) .
      2. Ongoing or active infection.
      3. Keratitis or onset of ulcerative keratitis.
      4. Other significant disease, mental illness or laboratory abnormalities that could affect the compliance of the patient on the protocol or investigator's judgement.
  11. Clinically significant, uncontrolled heart disease, including but not limited to:

      1. Abnormal QT interval on screening electrocardiogram (ECG), defined as the average value of triplicate QTcF>470ms.
      2. Have significant arrhythmias such as ventricular arrhythmia, supraventricular arrhythmia which could not be controlled by drugs, nodal arrhythmia and other cardiac arrhythmias which could not be controlled by drugs, Grade≥3 of Congestive heart failure by the New York Heart Association (NYHA).
      3. Any factors that increase the risk of QTc interval prolongation, such as hypokalemia, genetic long QT syndrome, taking drugs that causing the QT interval prolongation.
  12. Medical history of deep vein thrombosis or pulmonary embolism within 6 months prior to enrolment or any of the following: Myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Or bleeding tendencies or hypercoagulable coagulopathy within 6 months prior to first dose.
  13. Have active digestive system disease, or major gastrointestinal surgery which may significantly affect the taking or absorption of PLB1004(such as ulcerative lesions, uncontrollable nausea, vomiting, diarrhea, and malabsorption syndrome).
  14. History of hypersensitivity to active or inactive excipients of PLB1004 or drugs with a similar chemical structure of class to PLB1004.
  15. pregnant or nursing women.
  16. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
objective Response Rate (ORR) | 3 years
  To evaluate the Objective Response Rate（ORR）which is defined by IRC as the proportion of subjects with confirmed best overall response of complete response or partial response per RECIST v 1.1.

SECONDARY OUTCOMES:
objective Response Rate (ORR) | 3 years
  To evaluate the Overall Response Rate（ORR）which is defined by investigator as the proportion of subjects with confirmed best overall response of complete response or partial response per RECIST v 1.1.
Disease Control Rate ( DCR) | 3 years
  DCR is defined as the percentage of participants achieving complete or partial response or stable disease of at least 11 weeks as defined per RECIST v 1.1
Duration of Response (DOR) | 3 years
  DOR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first.
Progression-Free Survival (PFS) | 3 years
  PFS is defined as the time from the date the first dose until the date of objective disease progression or death by cause, whichever comes first, based on investigator review according to RECISTv1.1.
Overall Survival (OS) | 3 years
  OS is defined as the time from the date of the first dose until the date of death due to any cause.
Intracranial Overall Response Rate（ORR） | 3 years
  To evaluate the intracranial Overall Response Rate（ORR）which is defined by investigator as the proportion of subjects with Intracranial disease confirmed best overall response of complete response or partial response per RECIST v 1.1.
Intracranial Disease Control Rate (DCR) | 3 years
  Intracranial DCR is defined as the percentage of participants achieving Intracranial disease complete or partial response or stable disease of at least 11 weeks as defined per RECIST v 1.1.
Intracranial Disease Control Rate (DOR) | 3 years
  Intracranial DOR is defined as the time from the date of first documented response (CR or PR) until the date of Intracranial disease documented progression or death, whichever comes first.
Intracranial Progression-Free Survival (PFS) | 3 years
  Intracranial PFS is defined as the time from the date the first dose until the date of objective disease progression or death by cause, whichever comes first, based on investigator review according to RECISTv1.1.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | 2 years
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug assessed by CTCAE v5.0.
Incidence of abnormalities in Clinical Laboratory Assessments. | 2 years
  Number of participants with abnormalities in Clinical Laboratory tests（including serum chemistry and hematology） will be reported.
Incidence of abnormalities in Vital Signs. | 2 years
  Number of participants with abnormalities in vital signs(including temperature ,pulse/heart rate，and blood pressure) will be reported.
Area Under the Curve（AUC0-t）of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The AUC values are based on the plasma concentration-time profile (from time 0 to Time of the Last Quantifiable Concentration) of PLB1004. To characterize the pharmacokinetics of PLB1004.
Area Under the Curve（AUC0-∞）of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The AUC values are based on the plasma concentration-time profile (from time 0 to infinity) of PLB1004. To characterize the pharmacokinetics of PLB1004.
Maximum plasma concentration (Cmax) of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The Cmax values are based on the plasma concentration-time profile of PLB1004. To characterize the pharmacokinetics of PLB1004.
Time to maximum plasma concentration (Tmax) of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The Tmax values are based on the plasma concentration-time profile of PLB 1004.To characterize the pharmacokinetics of PLB1004.
Half-life time (t1/2) of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The t1/2 values are based on the terminal disposition Phase Half-life for PLB1004 and its Active Metabolites. To characterize the pharmacokinetics of PLB1004.
Apparent clearance (CL/F) of PLB1004 | Time Frame: Up to approximately 28 days; pre-dose and multiple time points post-dose
  The CL/F values are based on the apparent clearance after extravascular administration for PLB1004. To characterize the pharmacokinetics of PLB1004.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No